CLINICAL TRIAL: NCT04708834
Title: A Multicenter, Long-Term Open-Label Safety Study of Adjunctive Troriluzole in Subjects With Obsessive Compulsive Disorder
Brief Title: Long-term Safety Study of Adjunctive Troriluzole in Subjects With Obsessive Compulsive Disorder
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV4157-209
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive compulsive disorder; OCD; troriluzole; Biohaven
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Troriluzole (BHV-4157) (Experimental): 200 mg daily first 2 weeks, 280 daily following first 2 weeks
  Interventions: Drug: Troriluzole (BHV-4157)

INTERVENTIONS:
Drug: Troriluzole (BHV-4157) — 200 mg daily first 2 weeks, 280 daily following first 2 weeks

SUMMARY:
The purpose of the study is to evaluate the long term safety and tolerability of troriluzole as adjunctive therapy in subjects with obsessive compulsive disorder (OCD).

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible subjects are those subjects who complete study BHV4157-302 or BHV4157-303 and for whom the investigator believes open-label treatment offers an acceptable risk-benefit profile.
* Determined by the investigator to be medically stable at the week 10 visit of BHV4157-302 or BHV4157-303, as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing.
* It is required that all women of child-bearing potential (WOCBP) who are sexually active agree to use two methods of contraception for the duration of the study

Key Exclusion Criteria:

* Subjects who did not successfully complete 10 weeks of treatment in the BHV4157-302 or BHV4157-303 study.
* Acute suicidality or suicide attempt or self injurious behavior in the last 12 months.
* Patients who may have received a non-biological investigational agent in any clinical trial within 30 days or a biological agent within 90 days prior to entry, other than what was received in BHV4157-302 or BHV4157-303;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long term safety and tolerability of troriluzole as adjunctive therapy in subjects with OCD who have had an inadequate response to SSRI, clomipramine, venlafaxine or desvenfaxine treatment | Change from Baseline to week 240
  Percent change in treatment emergent adverse events, and clinical significant abnormalities in ECG's and lab values after Baseline.

CONTACTS AND LOCATIONS:
Locations (175):
- United States (147):
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - Alea Research, Phoenix, Arizona
  - NoeisisPharma, LLC, Phoenix, Arizona
  - Atria Clinical Research, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CITrials (Clinical Innovations), Bellflower, California
  - Southern California Research, LLC, Beverly Hills, California
  - Axiom Research, LLC, Colton, California
  - Global Clinical Trials, Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - WR-PRI, LLC (Encino), Encino, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Om Research LLC, Lancaster, California
  - Synergy Research San Diego, Lemon Grove, California
  - Alliance for Research, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - CalNeuro Research Group, Los Angeles, California
  - Clarity Clinical Research, Los Angeles, California
  - Pharmacology Research Institute (WR-PRI, LLC), Newport Beach, California
  - Pacific Research Partners, Oakland, California
  - North County Clinical Research, Oceanside, California
  - Excell Research, Inc, Oceanside, California
  - NRC Research Institute, Orange, California
  - Anderson Clinical Research, Redlands, California
  - CI Trials, Riverside, California
  - ACRC Studies, San Diego, California
  - Lumos Clinical Research Center, LLC, San Jose, California
  - National Research Institute, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Stanford University, Stanford, California
  - Collaborative Neuroscience Research, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Mountain View Clinical Research, Denver, Colorado
  - Institute of Living / Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Topaz Clinical Research, Apopka, Florida
  - Boca Raton Medical Institute, Boca Raton, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - CNS Research of Coral Springs, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - University of Florida Department of Psychiatry, Gainesville, Florida
  - Qway Research, LLC, Hialeah, Florida
  - Research in Miami Inc, Hialeah, Florida
  - Health Care Family Rehab & Research, Hialeah, Florida
  - Galiz Research, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Accel Research Sites (formerly Meridien Research), Lakeland, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Pharmaceutical Research Center, Inc., Lutz, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Meridien Research, Maitland, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Clintex Research, Miami, Florida
  - Sanchez Clinical Research Inc, Miami, Florida
  - Med-Care Research, Miami, Florida
  - FIRC, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Ezy Medical Research, Co., Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Pro-Care Research Center, Miami Gardens, Florida
  - South Florida Research Phase I-IV, Inc., Miami Springs, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Bayside Clinical Research, LLC, New Port Richey, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research, LLC, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - IMIC Inc, Palmetto Bay, Florida
  - MedBio Trials, Pembroke Pines, Florida
  - DMI Research, Pinellas Park, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Conquest Research LLC, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Renew Health Clinical Research, LLC, Snellville, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Uptown Research Institute, Chicago, Illinois
  - University of Chicago Department of Psychiatry & Behavioral Neuroscience, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - AMR-Baber Research, Inc, Naperville, Illinois
  - Collective Medical Research, Prairie Village, Kansas
  - Northern Light Acadia Hospital, Bangor, Maine
  - CBH Health, Gaithersburg, Maryland
  - Pharmasite Research, Inc., Pikesville, Maryland
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Sisu at RMG, Springfield, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Boeson Research, Missoula, Montana
  - Altea Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Bio Behavioral Institute, Great Neck, New York
  - Bioscience Research, LLC, Mount Kisco, New York
  - Hapworth Research, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Clinical Inquest Center, Ltd, Beavercreek, Ohio
  - NeuroScience Research Center, LLC., Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Central States Research, LLC, Tulsa, Oklahoma
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - BioBehavioral Research of Austin, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - DiscoveResearch, Inc. (DRI), Bryan, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Relaro Medical Trials, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Mt.Olympus Medical Research LLC, Missouri City, Texas
  - AIM Trials, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Woodstock Research Center, Woodstock, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - McMaster University, Hamilton Health Sciences, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - START Clinic for Mood and Anxiety Disorders, Toronto, Ontario
  - University of Toronto / Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
- Italy (5):
  - Institute of Neuroscience, University of Firenze, Florence
  - ASST FBF SACCO - Ospedale Universitario Luigi Sacco, Milan
  - University School of Medicine of Napoli Federico II, Naples
  - University of Pisa, Pisa
  - University of Turin - university hospital san luigi gonzaga, Turin
- Netherlands (2):
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- Spain (6):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Centro de Salud Mental La Corredoria, Oviedo
  - Centro de Salud San Juan, Salamanca
  - Hospital Álvaro Cunqueiro, Vigo
- United Kingdom (8):
  - MAC Clinical Research-Lancashire, Blackpool
  - Surrey and Borders Partnership NHS Foundation Trust, Chertsey
  - MAC Clinical Research -- Merseyside, Liverpool
  - South West London and St George's Mental Health NHS Trust Springfield University Hospital, London
  - MAC Clinical Research-Greater Manchester, Manchester
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester
  - Bioluminux Ltd, Milton Keynes
  - MAC Clinical Research-- South Yorkshire, Tankersley